CLINICAL TRIAL: NCT05365958
Title: Podcasting HIV Prevention Within African American Communities to Decrease New Infection
Brief Title: Podcasting HIV Prevention Within African American Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Chakema Carmack, Associate Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003312
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: HIV Prevention
Keywords: HIV Prevention; African Americans; Health Disparities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- African American Heterosexuals (Experimental)
  Interventions: Behavioral: HIV Podcast for Heterosexual African American Adults

INTERVENTIONS:
Behavioral: HIV Podcast for Heterosexual African American Adults — The video podcast will deliver HIV prevention messages using entertainment education and behavioral journalism, and film production techniques such as "talking head" video, interview, animations, & live-action skits. The research team will work closely with the production company in scripting the video vignettes and sequences, ensuring that video content reflects salient domains captured in the concept mapping research development phase of the study.

SUMMARY:
Given the continued impact of HIV among African Americans, there is still an urgent need to expand prevention efforts and HIV testing in African American communities. Heterosexual individuals may acquire and spread infection directly through heterosexual contact, bi-sexual sexual contact, and/or indirectly through homosexual sexual contact. Evidence-based interventions (EBIs) have been shown to increase consistent condom use, decrease sexual partners, and increase HIV testing; however, traditionally-implemented EBIs may not be accessible to communities given the resources and expertise needed to implement them. This project seeks to: 1) assess feasibility for the development of two theory- based, video podcast-delivered, HIV prevention interventions for self-identified heterosexual African American males and females; and 2) evaluate their feasibility & effectiveness (pilot). The investigators will develop the two (male and female) video podcasts that maintain the theoretical integrity of two established Centers for Disease Control evidence-based behavioral HIV prevention interventions. The assessment phase will consist of leveraging African American community stakeholders and experts in the development of the podcast content. The effectiveness phase will consist of broadcasting the podcasts for participants and evaluating psychosocial factors related to HIV prevention at 1 and 3 month follow-ups. This intervention is the first of its kind and has the potential to increase HIV protective behaviors in this hard-to-reach and medically underserved population. The resulting interventions are expected to be easily disseminated throughout the African American communities, with the potential to reduce HIV- related disparities within this population. This study will impact and advance the field by demonstrating feasibility and effectiveness for a novel mode of intervention engagement within HIV prevention science, serve as valuable preliminary data for a larger R01 trial, and foster HIV prevention awareness within the African American community.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American
* speak and read English
* 18 years old or older
* not currently or previously diagnosed with HIV

Exclusion Criteria:

• currently or previously diagnosed with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jacob's Home for Men, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Because this is a feasibility study with a low sample size, the data is preliminary and it is not certain that the data will be appropriate or useful for public dissemination.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 11, 2022 Recruitment at local community events, via social media, flyer distribution, churches.
Groups:
- African American Heterosexuals: Group participated in the pretest, intervention, & posttest/follow-up. (Single arm study)
Period: Overall Study
Arm/Group | African American Heterosexuals
Started | 128
Completed | 128
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | African American Heterosexuals
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: aggregate age] — Age (raw number)
  aggregate age | 36.2 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants] — This measure assessed binary biological gender: male/female
  Participants
    Female | 64
    Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 128
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The measure assesses U.S. Census-based terminology of "African American/Black" race. Self-identifying African American/Black was an eligibility criterion for this study; participants re-affirmed in the baseline measure that they were African American/Black.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 128
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 128
HIV-Knowledge Questionnaire [HIV KQ-14] [Mean (Standard Deviation); unit: scores] — 14-item HIV Knowledge Scale; 14 true/false items; summed for total scale score. Scores on the scale were the unit of measure. Scores range from 0 - 14. Higher scores indicate greater HIV knowledge; lower scores indicate less HIV knowledge.
  scores | 10.2 (2.2)
Psychosocial Aspects of HIV Prevention Behavior: Condom Use Self-Efficacy Subscale [Mean (Standard Deviation); unit: scores] — Researcher-created Condom Use Self-Efficacy scale (CUSE). The CUSE consists of 5-item that measure self-efficacy to use condoms. Each item response set was 1-Strongly disagree to 5-Strongly agree. Scale average ranged from 1 - 5. Higher scale scores indicate greater self-efficacy to use a condom during intercourse; Lower scale scores indicate lesser self-efficacy to use a condom during intercourse.
  scores | 3.0 (.7)
Psychosocial Aspects of HIV Prevention Behavior: Condom Use Intention Item [Mean (Standard Deviation); unit: scores] — Researcher-created scale with subscales of HIV-related attitudes, norms, efficacies, & intentions; adapted from previous scales. Reports results from the Condom Use Intention item. The condom use intention item consists of 1 item that measures intentions to use condoms. Item response set was 1-Strongly disagree to 5-Strongly agree, thus, scores on the scale ranged from 1 - 5. Higher scale scores indicate greater intentions to use a condoms; Lower scale scores indicate lower intentions to use a condom during intercourse.
  scores | 3.4 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Condom Use Self-Efficacy (From Baseline to 1 Month Follow-up)
Description: A change between baseline and 1 month regarding condom use self-efficacy scale scores.
  Results reflect mean difference and mean standard deviation in a repeated measures t-test analysis.
  The 5-item subscale scores were summed and averaged across participants, yielding an average scale score range of 1-5; higher scale values indicating greater self-efficacy to use condoms.
  Scale scores were assessed for participants immediately before the intervention and 1 month after the intervention. The method used was repeated measures t-test. The analysis reports the group average scale score and standard deviation for participants at 1 month followup.
Time Frame: To be measured immediately before film viewing (baseline) and at 1 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Heterosexuals
Number analyzed (Participants) | 128
score on a scale | 4.4 (.6)
Statistical Analysis 1: Comparison: African American Heterosexuals; Test type: Superiority; p < .001, Repeated Measures t-test of differences

2. Primary Outcome: Condom Use Intention Item (1 Month Followup)
Description: Uses the condom use intention item (average) of the measure. "I plan to use condoms the next time I have sex." Item was scaled from 1-strongly disagree to 5-strongly agree. Higher scale scores indicate greater intention to use a condom during intercourse; Lower scale scores indicate lesser intention to use a condom during intercourse.The item was summed across participants, separately for baseline and 1 month followup to yield a pretest group mean average (baseline) and a 1 month followup group mean average. The method used was repeated measures t-test, which tested group mean differences between baseline (pretest average) and 1 month followup average. The analysis reports the group average scale score and standard deviation for participants at 1 month followup.
Time Frame: To be measured 1 month after film viewing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Heterosexuals
Number analyzed (Participants) | 128
score on a scale | 4.1 (1.1)
Statistical Analysis 1: Comparison: African American Heterosexuals; Test type: Superiority; p < .001, Repeated Measures t-test of differences

3. Primary Outcome: HIV Test Intentions (Single Item)
Description: Uses a single item "I intend to obtain an HIV test within the next 2 months?" Item was scaled from 1-strongly disagree to 5-strongly agree. Higher scale scores indicate greater intention to acquire an HIV test; Lower scale scores indicate less intention to acquire an HIV test.The item scores were summed across participants, separately for baseline and 1 month followup to yield a pretest group mean average (baseline) and a 1 month followup group mean average. The method used was repeated measures t-test, which tested group mean differences between baseline (pretest average) and 1 month followup average. The analysis reports the group average scale score and standard deviation for participants at 1 month followup.
Time Frame: 1 month after film viewing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Heterosexuals
Number analyzed (Participants) | 128
score on a scale | 4.3 (.6)

4. Primary Outcome: Number of Participants With Who Have Obtained a HIV Test at 1 Month After Film Viewing
Description: To observe whether the film viewing influenced behavior of obtaining a HIV test at 1 month followup. Outcome was measured with a single item: "Have you obtained an HIV test (-you will not be required to disclose the results of this test)?" Item was scaled on a nominal scale of measurement as (0) No, (1) Maybe, and (2) Yes. A count of "Yes" (converted to percentage) was used as the primary outcome.
Time Frame: To be measured 1 month after film viewing
Measure: Count of Participants; unit: Participants
Arm/Group | African American Heterosexuals
Number analyzed (Participants) | 128
Participants | 18

5. Primary Outcome: Number of Participants With Who Have Obtained a HIV Test at 3 Months After Film Viewing
Description: To observe whether the film viewing influenced behavior of obtaining a HIV test at 3 month followup. Outcome was measured with a single item: "Have you obtained an HIV test (-you will not be required to disclose the results of this test)?" Item was scaled on a nominal scale of measurement as (0) No, (1) Maybe, and (2) Yes. A count of "Yes" (converted to percentage) was used as the primary outcome.
Time Frame: To be measured 3 months after film viewing
Measure: Count of Participants; unit: Participants
Arm/Group | African American Heterosexuals
Number analyzed (Participants) | 128
Participants | 53

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | African American Heterosexuals
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT05365958/Prot_SAP_000.pdf